CLINICAL TRIAL: NCT04628039
Title: Chronic Lung Disease and COVID-19: Understanding Severity, Recovery and Rehabilitation Needs (LAUREL Study)
Brief Title: Chronic Lung Disease and COVID-19: Understanding Severity, Recovery and Rehabilitation Needs
Acronym: LAUREL
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: F3666-R; 1I01RX003666-01 (NIH)
Record Dates: First submitted 2020-11-09; First posted 2020-11-13 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: COVID-19; Chronic Lung Diseases
Keywords: Chronic Lung Disease; COVID-19; Rehabilitation; Veterans; SARS-CoV-2; COPD
MeSH Terms: conditions — COVID-19; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- COVID Positive: Veterans aged 18 years or older who have a positive SARS-CoV-2 diagnosis (confirmed or presumptive) or who have been discharged home within 2 weeks to 1 year of diagnosis
- COVID Negative and Lower Respiratory Tract Infection (LRTI): Veterans aged 18 years or older with a negative SARS-CoV-2 test (PCR and/or antigen test) and diagnosis of LRTI after discharge home or after diagnosis if not hospitalized

SUMMARY:
This is study is comprised of three approaches. First, the investigators will conduct a retrospective cohort study to determine factors associated with COVID-19 severity and complications and understand COVID-19 outcomes, including all-cause mortality, post-discharge events, and impacts of rehabilitation services (third aim). The second aim is a mixed-method study and follows COVID-19 patients with repeated surveys to determine patient-reported functional outcomes, health recovery, and rehabilitation needs after COVID-19. The investigators will recruit patients and their informal caregivers for interviews to assess their function and rehabilitation needs.

DETAILED DESCRIPTION:
The long-term consequences of COVID 19 are not well understood, particularly in the Veteran population. This study will describe and quantify the long-term consequences of COVID-19, including impairment in physical and psychosocial function and health-related quality of life. Additionally, it will determine the impact of chronic lung disease (CLD) and other comorbidities on severity and recovery after COVID-19 infection and the association of social determinants of health with severity and recovery.

Initially, a retrospective national cohort of VA patients who test positive with SARS2 will be identified. Baseline clinical history will be analyzed with outcomes that include severity of COVID 19, all-cause mortality, and post-discharge events.

Subsequently, a mixed methods, prospective cohort study will include both qualitative (interview) and quantitative components (surveys). The investigators will identify patients with COVID-19 and recruited for qualitative interviews following hospital discharge or diagnosis. Patient caregivers will also be eligible to participate in study interviews. Interviews will occur once at various times ranging 2 weeks to 1 year since a patient's COVID-19 diagnosis. Surveys will be completed at 3 time points, 2-8 weeks after diagnosis or discharge to home, and then 6 months and 12 months later. Surveys will include the EQ-5D-5L profile for health-related quality of life, and the WHODAS 2.0 score for a global assessment of overall physical and psychosocial function. Investigators will also identify a comparator cohort of patients who have been diagnosed with lower respiratory tract infection (LRTI) in the setting of a negative COVID-19 test. Surveys will be administered at the same interval and analysis will determine if COVID-19 has different and more severe health impacts than other causes of lower respiratory tract infection.

ELIGIBILITY:
Inclusion Criteria:

* (Patients in COVID-19 cohort) VA patients diagnosed with COVID-19 through a positive PCR (Polymerase Chain Reaction) or antigen SARS-CoV-2 test conducted in VA
* (Caregivers) Providing caregiving to VA patients diagnosed with COVID-19
* (Patients in LRTI cohort) VA patients diagnosed with LRTI and tested negative for COVID-19 (through PCR and/or antigen test)

Exclusion Criteria:

* Cognitive limitations that preclude the ability to communicate and obtain informed consent
* Language barriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans aged 18 years or older who have a positive SARS-CoV-2 diagnosis (confirmed or presumptive) or who have been discharged home within 2 weeks to 1 year of diagnosis. Those who do not speak English or have cognitive limitations that preclude the ability to communicate and obtain informed consent will be excluded
Sampling Method: Probability Sample
Enrollment: 622 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
EuroQol 5 Dimension 5 Level (EQ-5D-5L) visual analog score | Change in score from 3-8 weeks (after diagnosis or discharge to home) to months 6 and 12
  Profile for health-related quality of life. The investigators will summarize this measure with a visual analog score (VAS). The VAS ranges from 0 to 100mm (where 0="the worst health you can imagine"; 100="the best health you can imagine").
WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) | Change in score from 3-8 weeks (after diagnosis or discharge to home) to months 6 and 12
  Global assessment of overall physical and psychosocial function. The overall score for disability will be calculated using item-response-theory (IRT) based scoring. This scale ranges from 0 to 100 (where 0 = no disability; 100 = full disability).
EuroQol 5 Dimension 5 Level (EQ-5D-5L) overall utility index | Change in score from 3-8 weeks (after diagnosis or discharge to home) to months 6 and 12
  Profile for health-related quality of life. We will summarize this measure with an overall utility index. The utility index ranges from less than 0 to 1(where <0="worse than death";1=full health).

CONTACTS AND LOCATIONS:
Overall Officials: Kristina A Crothers, MD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turner AP, Adams SV, Hawkins E, Fan VS, Nikzad R, Kundzins JR, Crothers K. Alcohol Use and COVID-19 Outcomes. Chest. 2025 Sep;168(3):589-601. doi: 10.1016/j.chest.2025.05.039. Epub 2025 Jun 10. PMID 40505809
- [Derived] Petrova VV, Turner AP, Simons C, Kamiab NA, Crothers K, Sayre GG. Veterans' Experiences with COVID-19 and How Providers Can Shape Care and Perception with Empathy. J Gen Intern Med. 2025 May 15. doi: 10.1007/s11606-025-09557-9. Online ahead of print. PMID 40375042
- [Derived] Crothers K, Adams SV, Turner AP, Batten L, Nikzad R, Kundzins JR, Fan VS. COVID-19 Severity and Mortality in Veterans with Chronic Lung Disease. Ann Am Thorac Soc. 2024 Jul;21(7):1034-1043. doi: 10.1513/AnnalsATS.202311-974OC. PMID 38530061

DOCUMENTS (1):
  • Informed Consent Form (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT04628039/ICF_000.pdf